CLINICAL TRIAL: NCT05479175
Title: Evaluation the Effect of Using Preoperative Ibuprofen Versus Low Level Laser Therapy on Inferior Alveolar Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Assoc.Prof, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/15.12.2021
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain
Keywords: Root canal; anesthesia; inferior alveolar nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Group 1: Ibuprofen 600 mg will be given to the patient one hour before starting root canal treatment.
  Group 2: Low-level laser therapy will be applied with an 810 nm wavelength diode laser device for 30 seconds in the area of mesial root and 30 seconds in the area of distal root , total of 60 seconds.
  Group 3: Placebo, will be explained to the patients that laser treatment will be applied as in group 2, but laser will not be activated.
  Group 4: Control, routine root canal treatment will be done. No medication or laser will be applied before the treatment procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ibuprofen (Active Comparator): Ibuprofen 600 mg will be given to the patient one hour before starting root canal treatment.
  Interventions: Drug: Ibuprofen
- Diode laser (Active Comparator): Low-level laser therapy will be applied with an 810 nm wavelength diode laser device for 30 seconds in the area of mesial root and 30 seconds in the area of distal root , total of 60 seconds.
  Interventions: Device: Diode laser
- Nonactive Diode laser (Active Comparator): Placebo, will be explained to the patients that laser treatment will be applied as in group 2, but laser will not be activated.
  Interventions: Device: Nonactive Diode laser
- Control (No Intervention): Control, routine root canal treatment will be done. No medication or laser will be applied before the treatment procedure.

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen
  Arms: Ibuprofen
Device: Diode laser — Diode laser
  Arms: Diode laser
Device: Nonactive Diode laser — Nonactive Diode laser
  Arms: Nonactive Diode laser

SUMMARY:
Acute apical periodontitis (AAP) is an inflammatory condition of the periapical tissues of the periodontium, usually resulting from irreversible pulpitis and pulpal necrosis. Patients with AAP often have moderate to severe pain, which results in the need for emergency treatment. Patients with AAP usually present with dull, throbbing, constant pain; absence of swelling; a negative or delayed positive result on vitality testing; absence of thermal sensitivity of the tooth; and pain on biting or percussion.The treatment of these teeth is root canal treatment. Pain control during root canal treatment is essential for several reasons. First, patients desire and expect that their treatment should be free of discomfort. Second, good intra-operative pain control helps to reduce post-operative pain and simplifies its management. Third, patients will be reluctant to have further root canal treatment in the future if they have had a bad experience as a result of pain during treatment. Hence, pain-free treatment should be every dentist's aim. The amount of pain experienced during treatment is related to the condition being treated teeth with irreversible pulpitis and acute apical periodontitis were significantly associated with more treatment pain than devital teeth and infected canals with apical periodontitis.In another study, molars and teeth with irreversible pulpitis had more intra-operative pain than single-rooted teeth and devital teeth, infected root canals. Local anesthesia is the most common method used for pain control during root canal treatment. However, other strategies can also be employed in some cases such as pre-treatment anti-inflammatory systemic medications, and methods to reduce discomfort associated with injections. The use of pre-operative medication reduce pain and inflammation at the treatment site. Several studies have been performed to investigate the effectiveness of this approach using a variety of drugs such as benzodiazepines, NSAIDs and corticosteroids. The concept of using NSAIDs and corticosteroids as premedication is largely based on reducing the amount of prostaglandin in the inflamed pulp. There have been conflicting results reported for the use of ibuprofen premedication with some studies reporting an increased success rate for local anaesthesia,while others have reported no effects compared with placebo.

Recently, low level laser therapy has been used in dentistry for a range of treatments, including reduction of orthodontic pain, symptomatic oral lichen planus cases, healing of maxillofacial defects and prophylaxis of stomatitis. LLLT has begun to be used in endodontic treatments due to its ability to increase wound healing, its role in root canal disinfection, its role in reducing pain and its very limited side effects. However, the pain reduction mechanism of LLLT is not fully understood.

DETAILED DESCRIPTION:
The study is to be carried out in 76 medically free patients, aged 18-50 years, who were diagnosed in Van Yuzuncu Yıl University, Faculty of Dentistry, Department of Endodontic, The number of patient was calculated in the G* Power 3.1 software. In this study cohen criteria was used. Taking effect size 0.40, alpha = 0.05, and power = 0.80, the minimum number of patients was determined as 76.

Lower first and second molars (36,37,46,47) diagnosed with acute apical periodontitis will be included in the study as an experimental group. Patients with periapical lesions and open apex teeth will not be included in the study group. Preoperative pain degree will be determined using Visual analogue scale (VAS) test. Patients will be randomly divided into 4 groups.

Group 1: Ibuprofen 600mg will be given to the patient one hour before starting root canal treatment Group 2: Low-level laser therapy will be applied with an 810 nm wavelength diode laser device for 30 seconds in the area of mesial root and 30 seconds in the area of distal root , total of 60 seconds .

Group 3: Placebo, will be explained to the patients that laser treatment will be applied as in group 2, but laser will not be activated.

Group 4: Control, routine root canal treatment will be done. No medication or laser will be applied before the treatment procedure.

After applying 2 ml ultracain DS forte local anesthesia access cavity will be opened. The working length will be determined using the apex locator by placing a K file #15 into the root canals until the apical constriction. The shaping process of the root canals will be done by ProTaperNext files up to the X3 as standard in all patients. 2 ml of 5.25% NaOCl irrigation solution will be applied after each file. A 2 ml dental injector with a 27 gauge dental needle will be used and The tip of the needles will be adjusted to be 2mm shorter than the working length. After complete the cleaning and shaping process, the root canals will be filled with gutta-percha and ADSEAL resin sealer using the lateral condensation technique. After complete the root canal treatment, the level of pain experienced by the patients during the treatment will be determined using the visual analogue scale (VAS) test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 50 years
* Mandibular molar teeth that were diagnosed with acute apical periodontitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with calcified canals
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS Scale | up to 2 hours
  PP will be assessed with a VAS after endodontic treatment. The VAS consisted of a 100-mm hor- izontal ruler with marks every 10 mm and no numbers except a 0 at the first part of the scale and a 10 in the last part of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Özlek, PhD, Study Director — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasanna N, Subbarao CV, Gutmann JL. The efficacy of pre-operative oral medication of lornoxicam and diclofenac potassium on the success of inferior alveolar nerve block in patients with irreversible pulpitis: a double-blind, randomised controlled clinical trial. Int Endod J. 2011 Apr;44(4):330-6. doi: 10.1111/j.1365-2591.2010.01833.x. PMID 21692235